CLINICAL TRIAL: NCT07312318
Title: DeVelopment of an Artificial Intelligence-Driven Dynamic Prediction and Precision Stratification System for Coronary Non-Target LesIon ProgressiON After Percutaneous Coronary Intervention: A Multimodal Data-Enabled Multicenter Cohort Study in China
Brief Title: AI-Driven Dynamic Prediction of Non-Target Lesion Progression After PCI: A Chinese Multicenter Cohort Study
Acronym: VISION-PCI
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Fang Wang, Associate Professor of Cardiology Department, China-Japan Friendship Hospital
Other Study IDs: 2025-NHLHCRF-PY-07
Record Dates: First submitted 2025-12-03; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Coronary Heart Disease (CHD)
Keywords: Artificial Intelligence; Non-Target LesIon Progression; Percutaneous Coronary Intervention; coronary heart disease
MeSH Terms: conditions — Coronary Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Biospecimen Retention: Samples Without DNA — Collect 4 ml of fasting peripheral venous blood from enrolled patients. Fasting should commence at 22:00 the day before blood collection. The blood should be placed in EDTA anticoagulant tubes. Within 2 hours after blood collection, plasma should be separated and stored for subsequent lipidomic analysis. This involves centrifuging at 3000 rpm for 10 minutes to separate the plasma. Transfer the upper layer of plasma into 200 ul/1.5 ml EP tubes, then store at
  -80°C for preservation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: percutaneous coronary intervention — Percutaneous coronary intervention (PCI) represents a cornerstone therapeutic approach for coronary artery disease. This minimally invasive procedure involves vascular access typically through the radial or femoral artery, enabling the navigation of catheters and specialized devices to the culprit coronary lesion. The primary objective is to restore optimal coronary blood flow by addressing the obstructive lesion. The intervention encompasses various techniques including balloon angioplasty, stent implantation, and adjunctive procedures such as coronary atherectomy and thrombus aspiration when clinically indicated.

SUMMARY:
Coronary artery disease remains a leading cause of global mortality. Although percutaneous coronary intervention (PCI) improves patient outcomes, the long-term risk of major adverse cardiovascular events (MACE) driven by the progression of non-target lesions (NTLs) remains substantial and continues to increase, while current risk stratification tools remain inadequate for predicting NTL progression. This multicenter cohort study aims to develop an artificial intelligence (AI)-driven system for the dynamic prediction and precision stratification of NTL progression after PCI. Utilizing comprehensive multimodal data from 52,577 Chinese patients-including clinical profiles, multi-omics blood biomarkers, and coronary imaging-the research pursues three primary objectives: (1) to identify and validate 2-3 specific biomarkers for NTL progression risk using multi-omics approaches; (2) to construct an integrated risk assessment and early-warning system by applying machine learning to multimodal data for predicting NTL progression and MACE; and (3) to establish metabolic and imaging-based subtypes to create a precision management system that optimizes secondary prevention strategies by identifying specific high-risk populations. This study is expected to provide a novel tool for accurate identification of high-risk patients and personalized post-PCI management, ultimately aiming to improve long-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. Scheduled for or having undergone PCI;
3. Baseline plasma sample obtainable;
4. Informed consent obtained

Exclusion Criteria:

1. Pregnancy or lactation;
2. Severe hepatic or renal dysfunction;
3. Active autoimmune disease;
4. Missing critical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study integrates three dedicated Chinese cohorts of post-PCI coronary artery disease patients, comprising two cohorts provided by the National Population Health Data Center and one consecutive cohort recruited from the Department of Cardiology at China-Japan Friendship Hospital.
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of NTL progression-related myocardial infarction or revascularization | 12 month follow-up
  1. NTL progression-related myocardial infarction was defined in accordance with the fourth universal definition of myocardial infarction due to any segment of the nontarget vessel or lesion.
  2. NTL progression-related revascularization was defined as revascularization driven by angina or ischemia, either PCI or CABG, of any segment of the nontarget vessel or lesion.

SECONDARY OUTCOMES:
Qualitative data on NTL progression | 12 month follow-up
  The following conditions are defined as NTL progression: (1) NCL stenosis ≥50% at baseline PCI with ≥10% NCL progression at angiographic follow-up; (2) NCL stenosis <50% at baseline PCI with ≥30% NCL progression at angiographic follow-up; (3) NCL progression ≥30% without NCL at baseline PCI; (4) NCL progression to complete occlusion. Quantitative data for NTL progression (QCA) are obtained by analyzing coronary angiographic images to determine lesion progression.
Quantitative data on NTL progression | 12 month follow-up
  QCA analyzes coronary angiography images to determine the progression of lesions: Coronary angiography was evaluated by two independent cardiologists who were unaware of all other clinical data of the patients, using the MEDCON TCS QCA software. First, the edges of the contrast-enhanced vessels were delineated using an automatic edge detection algorithm. After identifying the starting and ending points on the enhanced coronary images, a vascular path was created. Subsequently, the vessel contour was drawn along the path. The path and vessel contour were automatically determined based on contrast density, with occasional manual editing required by the analysts. Measured variables included minimum lumen diameter and degree of lumen stenosis (minimum lumen diameter/adjacent contrast vessel diameter).
NTL progression-related myocardial infarction | 12 month follow-up
  NTL progression-related myocardial infarction was defined in accordance with the fourth universal definition of myocardial infarction due to any segment of the nontarget vessel or lesion.
NTL progression-related revascularization | 12 month follow-up
  NTL progression-related revascularization was defined as revascularization driven by angina or ischemia, either PCI or CABG, of any segment of the nontarget vessel or lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Wang, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided